CLINICAL TRIAL: NCT02134327
Title: Effect of Dexmedetomidine Versus Midazolam Versus a Combination of the Two as a Premedication for Children Undergoing Bilateral Myringotomy Tube Insertion: A Randomized, Blinded Study
Brief Title: Effect of Dexmedetomidine Versus Midazolam Versus a Combination of the Two as a Premedication for Children Undergoing Bilateral Myringotomy Tube Insertion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decided not to proceed
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JB004-1
Record Dates: First submitted 2014-05-01; First posted 2014-05-09 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Pre Operative Sedation; Mask Acceptance; Post Operative Delerium
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Premedication with Midazolam (Experimental)
  Interventions: Drug: Combination of Dexmedetomidine with Midazolam

INTERVENTIONS:
Drug: Combination of Dexmedetomidine with Midazolam

SUMMARY:
Following an obtained written consent, a child presenting for ear tube surgery will be randomized into one of three groups for receiving a premedication. One group will be the current therapy with midazolam, another group will be another drug dexmedetomidine, and the third group will be a combination of midazolam plus dexmedetomidine. Observers in the study (the investigators fellow and advance practice nurse) will not know which group each patient belongs, and will then make three separate assessments: preoperative sedation, mask acceptance, and postoperative delirium.

Mask acceptance: Induction of anesthesia, or the beginning of the process for the patient to fall asleep and lose consciousness, involves placing a mask over there face, specifically the nose and mouth. The mask is connected to their anesthesia machine via tubing, or a circuit, through which their anesthetic gases flow. Some children fight the mask as it can be seen as new and frightening. Other children, sometimes depending on how sedated they are after receiving a premedication, do not fear the mask on their face and do not resist induction. How well or easily this happens can be described as "mask acceptance." Postoperative delirium can be seen in patients of any age or after any surgery and can be better defined as a mental disturbance during the recovery from general anesthesia consisting of hallucinations, delusions, and confusion manifested by moaning, restlessness, involuntary physical activity, and thrashing about in bed. It has been considered a common postanesthetic problem in children and adults since 1960.

Each patient will then have a set of numbers for each scale; following conclusion of the study the investigators will be able see which drug each patient received and statistical analysis can be completed. The investigators goal is to see if there is any difference in any of the scales depending which medication was administered. The scales to be utilized include the pre-operative sedation scale, the mask acceptance scale, and the pediatric emergence delirium scale.

DETAILED DESCRIPTION:
Children presenting for ear tube surgery (bilateral myringotomy and ventilating tube insertion) often suffer from postoperative delirium in the recovery room. It has been hypothesized this may be a result or side effect of a premedication, midazolam. Midazolam is frequently administered to children preoperatively as a means of decreasing separation anxiety. An alternative medication, dexmedetomidine, is sometimes used as an alternative to midazolam and has also been effective in treating postoperative delirium. In this study the investigators would like to see if there is in fact a measurable difference between children receiving the standard midazolam or dexmedetomidine.

Patients would be randomized into one of three groups (versed alone, dexmedetomidine alone, or a combination). Patients included would be those presenting for BMT surgery who are an ASA physical status 1 or 2, not falling into any exclusion criteria.

Exclusion criteria would be patients with vital signs outside the normal limits as documented under the research plan. Also to be excluded are those patients with known genetic abnormalities predisposing to a derangement in hemodynamics or challenging airway.

The anesthesiologists listed as team members are the ones who are involved with this study and would be responsible for providing a standard anesthetic (same technique with inhalational anesthetic agents and intraoperative pain management) so no other variability would need to be taken into consideration for assessment in the recovery room. The investigators researchers, both anesthesiologists and observers will be blinded during the study. The pharmacy will have a list of patients who have consented, and then will randomly allocate them into one of the three groups. Only for analysis will the investigators (myself as the PI and other members) know which patient received which drug or combination. Also, by having the same team members performing assessment of each of the three parameters (1. Pre-op sedation scale, 2. Mask acceptance score, and 3. Post operative emergence delirium scale), there would be good reliability. A briefing session will be performed prior to the study's commencement showing pictures to the reviewers so there can be an agreed upon assessment. The MOASS or pre-operative sedation scale as well as the mask acceptance and PAED scale have been utilized and validated in previous studies (10), while the mask acceptance scale has been successfully utilized as well (11, 12, 13). The investigators goal is to decrease variability by having only two members make observations.

DESCRIPTION IN LAYMEN TERMS. Please summarize this study in less than 10 sentences. Use language an informed non-scientist can understand. Please complete within space below.

Following an obtained written consent, a child presenting for ear tube surgery will be randomized into one of three groups for receiving a premedication. One group will be the current therapy with midazolam, another group will be another drug dexmedetomidine, and the third group will be a combination of midazolam plus dexmedetomidine. Observers in the study (the investigators fellow and advance practice nurse) will not know which group each patient belongs, and will then make three separate assessments: preoperative sedation, mask acceptance, and postoperative delirium.

Mask acceptance: Induction of anesthesia, or the beginning of the process for the patient to fall asleep and lose consciousness, involves placing a mask over there face, specifically the nose and mouth. The mask is connected to their anesthesia machine via tubing, or a circuit, through which their anesthetic gases flow. Some children fight the mask as it can be seen as new and frightening. Other children, sometimes depending on how sedated they are after receiving a premedication, do not fear the mask on their face and do not resist induction. How well or easily this happens can be described as "mask acceptance." Postoperative delirium can be seen in patients of any age or after any surgery and can be better defined as a mental disturbance during the recovery from general anesthesia consisting of hallucinations, delusions, and confusion manifested by moaning, restlessness, involuntary physical activity, and thrashing about in bed. It has been considered a common postanesthetic problem in children and adults since 1960.

Each patient will then have a set of numbers for each scale; following conclusion of the study the investigators will be able see which drug each patient received and statistical analysis can be completed. The investigators goal is to see if there is any difference in any of the scales depending which medication was administered. The scales to be utilized include the pre-operative sedation scale, the mask acceptance scale, and the pediatric emergence delirium scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 mo-4 years
* ASA classification 1 or 2
* Vital signs, namely heart rate and blood pressure within the normal range for each patient's age group

Exclusion Criteria:

* Known allergies to midazolam or dexmedetomidine
* Baseline vitals outside the range listed above
* Personal or family history of malignant hyperthermia
* Genetic abnormalities predisposing to altered hemodynamics or difficult airway
* ASA physical status 3 or greater
* Known cardiac abnormalities

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Post operative anesthesia emergence delerium scale | From beginning of when patient receives medication for assessing preoperative sedation to recovery room when postoperative delerium is assessed. This whole process takes approximately 90 minutes.
  The primary outcome will be which group of subjects have different PAED or emergence derlium scale scores.

CONTACTS AND LOCATIONS:
Locations (1):
- A.I. Dupont Hospital for Children, Wilmington, Delaware, United States